CLINICAL TRIAL: NCT06949787
Title: Comparison of Spontaneous Onset of Labor and Vaginal Delivery in Post-date Primigravida Undergoing Sweeping of Membranes Versus Expectant Management
Brief Title: To Compare Sweeping of Membranes Versus Expectant Management for Spontaneous Onset of Labor and Vaginal Delivery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DrAyeshaCMHAttock
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Post-Term Pregnancy
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Membrane sweeping group (Experimental): Participants in the membranes sweeping group will receive membrane sweeping. If labor will not initiate within 48 hours, the procedure will be repeated up to a maximum of three times at 48-hour intervals.
  Interventions: Procedure: Membrane sweeping
- Expectant management group (No Intervention): Women in the expectant management group will receive no mechanical intervention, and these women will be monitored according to the standard protocol until spontaneous labor onset or labor induction will be deemed necessary.

INTERVENTIONS:
Procedure: Membrane sweeping — Participants in the membranes sweeping group will receive membrane sweeping. If labor will not initiate within 48 hours, the procedure will be repeated up to a maximum of three times at 48-hour intervals.
  Arms: Membrane sweeping group

SUMMARY:
The study is planned to fill the gaps regarding the effectiveness of sweeping of membranes versus expectant management in terms of spontaneous onset of labor and vaginal delivery in post-date primigravida.

DETAILED DESCRIPTION:
This study is important as it provides localized data on the effectiveness and practicality of membrane sweeping in a low-resource setting, which is underrepresented in current literature. Potential benefits of this research may include reduced need for formal labor induction, lower healthcare costs, and improved maternal and neonatal outcomes. The findings may enhance clinical practices by offering an evidence-based, patient-friendly approach to managing postdate pregnancies, particularly in resource-limited settings where induction facilities are constrained.

ELIGIBILITY:
Inclusion Criteria:

* Primigravid women
* Aged between 18 and 40 years
* Gestational age ≥40 weeks, confirmed by ultrasound or early dating scan
* Singleton pregnancies
* Cephalic presentation

Exclusion Criteria:

* Multiple gestations
* Fetal distress or anomalies detected on ultrasound
* Contraindications to vaginal delivery (e.g., placenta previa, previous uterine surgery)
* Previous uterine scar

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Spontaneous onset of labor and vaginal delivery | 6 days
  The occurrence of regular uterine contractions (contractions occurring every 3-5 minutes, each lasting 30-60 seconds, and progressively increasing in intensity) leading to cervical changes without any form of labor induction will mark the achievement of spontaneous onset of labor.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Ashraf, Principal Investigator — Combined military hospital, Attock, Pakistan; Tahir Ashraf, FCPS, Study Director — Combined military hospital, Attock, Pakistan
Locations (1):
- Combined Military Hospital, Attock, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
If a reasonable request is made, the data can be shared.